CLINICAL TRIAL: NCT04676373
Title: A Single Arm, Prospective, Open-label, Multi-center Study to Evaluate Efficacy and Safety in Chinese Patients With Late Onset Pompe Disease With Alglucosidase Alfa Treatment
Brief Title: Study to Evaluate Efficacy and Safety in Chinese Patients With Late Onset Pompe Disease With Alglucosidase Alfa Treatmen
Acronym: APOLLO-LOPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALGMYL09010; U1111-1238-1267 (Other: UTN); LPS15677 (Other: Sanofi Identifier); 2024-000461-24 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alglucosidase Alfa (Experimental): A dose of 20 mg/kg body weight once every 2 weeks for a minimum of 52 weeks
  Interventions: Drug: ALGLUCOSIDASE ALFA

INTERVENTIONS:
Drug: ALGLUCOSIDASE ALFA — Pharmaceutical form:solution for infusion
  Route of administration: intravenous
  Other Names: MYOZYME

SUMMARY:
Primary Objective:

To evaluate the effect of one-year Alglucosidase alfa treatment on motor function [Six-minute walk test (6MWT) and lung function predicted Forced vital capacity (FVC)] among Chinese Late Onset Pompe Disease patients above 5 years old.

To evaluate the safety of Myozyme 20mg/kg, IV biweekly in Chinese LOPD patients above 3 years old.

Secondary Objective:

To evaluate the effect of one-year treatment with Alglucosidase alfa on improvement of manual muscle test (MMT), Maximal inspiratory and expiratory pressure (MIP and MEP)], Quick Motor Function Test scores, and health-related quality of life (SF-12) among LOPD patients over 5 years old.

DETAILED DESCRIPTION:
Study duration per participants is approximatively 56 weeks including a 52-week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Patients (or and patient's legal guardian) must provide written informed consent prior to any study-related procedures
* The patient must be ≥ 3 years of age at the time of enrollment.

  1. For patient ≥ 3-year and < 5-year old: must be able to walk 10 meters or climb 4-step stairs independently.
  2. For patients ≥5-year old

  i. Must be able to ambulate 40 meters in 6 minutes without assistance ii. Must be able to successfully perform repeated forced vital capacity (VC) measurements in upright position of ≥ 30% predicted and ≤85% predicted.
* The patient has confirmed Pompe's Disease with at least 2 of the following condition,

  1. GAA enzyme deficiency from any tissue source.
  2. 2 confirmed GAA gene mutations.
  3. muscle pathology meet the diagnosis of Pompe disease.
* The patient (and patient's legal guardian if patient is legally minor as defined by local regulation) must have the ability to comply with the clinical protocol.
* The patient, if female and of childbearing potential, must have a negative pregnancy test (beta-human chorionic gonadotropin) at baseline.

Exclusion criteria:

* Use of invasive ventilatory support (Invasive ventilation is defined as any form of ventilatory support applied with the use of an endotracheal tube.)
* Use of non-invasive ventilatory support while awake and in an upright position. (Non-invasive ventilation is defined as any form of ventilatory support applied without the use of an endotracheal tube.)
* Previously treated with Enzyme Replacement Treatment.
* A Female patient of childbearing potential with a positive pregnancy test.
* Wheelchair dependent.
* The patient has a major congenital anomaly.
* The patient has a medical condition, serious intercurrent illness, or other extenuating circumstance, in the opinion of the Investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities.
* The patients with ≥5-year old are unable to ambulate 40 meters without assistance or unable to successfully perform repeated FVC of >30% and <85% predicted (upright).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Six-minute walk test (6MWT) for the patients ≥5-year old | Baseline to 12 months
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Change from baseline in percent predicted forced vital capacity (%FVC) in upright position for the patients ≥5-year old | Baseline to 12 months
  The measurements of pulmonary function and respiratory strength including FVC, MEP and MIP use a pneumograph or the spirometry system with the patient in upright seated and supine positions, according to American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
Number of participants with adverse events Number of AEs | From signing the ICF to the 30th day after the last dosage of the study medications
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from baseline in maximal inspiratory pressure (MIP) in upright position for the patients ≥5-year old | Week 52
  The measurements of pulmonary function and respiratory strength including FVC, MEP and MIP use a pneumograph or the spirometry system with the patient in upright seated and supine positions, according to American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
Change from baseline in maximal expiratory pressure (MEP) in upright position for the patients ≥5-year old | Week 52
  The measurements of pulmonary function and respiratory strength including FVC, MEP and MIP use a pneumograph or the spirometry system with the patient in upright seated and supine positions, according to American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
Change from baseline in manual muscle test (MMT) for deltoid muscle, quadriceps femoris, iliopsoas, neck stretch flexor for the patients ≥5-year old | Week 52
  MMT has been reported most often as a summary score of a total number of proximal, distal, and axial muscle groups tested bilaterally or as a proximal score that sums a number of proximal muscle groups from the upper and lower extremities.
Change from baseline in Quick Motor Function Test scores for the patients ≥5-year old | Week 52
  The Quick Motor Function Test is a reliable and valid test for assessing motor function in patients with Pompe's disease.
Change from baseline in Quick Motor Function Test scores for the patients ≥5-year old | Week 52
  The 12-Item Short Form Health Survey (SF-12) was developed for the Medical Outcomes evaluation of patients with chronic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ALGMYL09010 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25216&tenant=MT_SNY_9011